CLINICAL TRIAL: NCT06328348
Title: Assessing the Synergistic Effects of Black Cohosh, Soy Isoflavones, and SDG Lignans (Soloways TM) on Menopausal Symptoms: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: Assessing the Synergistic Effects of Black Cohosh, Soy Isoflavones, and SDG Lignans (Soloways TM) on Menopausal Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S.LAB (SOLOWAYS) (Other)
Collaborators: Center of New Medical Technologies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SW010
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Menopause Symptoms
Keywords: Postmenopausal women; Menopause Rating Scale; supplementation; lignans
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- supplementation group (Experimental)
  Interventions: Dietary Supplement: supplementation
- placebo group (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: supplementation — group receiving a course of Black Cohosh, Soy Isoflavones, and SDG Lignans
  Arms: supplementation group
Other: placebo — placebo
  Arms: placebo group

SUMMARY:
This clinical trial aimed to evaluate the effectiveness of a combination of Black Cohosh, Soy Isoflavones, and SDG Lignans compared to a placebo in reducing menopausal symptoms in postmenopausal women aged 45-60 years. The study was meticulously designed to be a randomized, double-blind, parallel-group trial, ensuring rigorous scientific standards and participant confidentiality. It received ethical approval and adhered to the Declaration of Helsinki guidelines. Participants were carefully selected based on specific inclusion and exclusion criteria to maintain the study's integrity and relevance to the target population.

The trial involved 96 eligible women from the Center for New Medical Technologies registry in Novosibirsk, Russia, divided into two groups through a computer-generated random sequence. One group received the active supplements, while the other received a placebo, with both groups and researchers blinded to the assignments. The supplements and placebos were produced to be indistinguishable in appearance, with dosages designed to maximize absorption and efficacy while minimizing side effects. The primary endpoint was the change in Menopause Rating Scale (MRS) scores, with secondary outcomes focusing on adverse symptoms and key hormonal changes.

The study's design also included measures to ensure adherence and minimize bias, such as drug container returns and daily reminders. The involvement of S.Lab (Soloways) was limited to manufacturing the supplements, with the research conducted independently to avoid commercial influence. The sample size calculation indicated that 48 participants per group would provide adequate power to detect significant differences in menopausal symptom reduction, aiming for a high level of confidence and statistical power.

ELIGIBILITY:
Inclusion Criteria:

* Time since menopause less than 10 years
* Natural menopause confirmed
* Abstainers from smoking and alcohol consumption
* Normal thyroid function tests and lipid profiles
* Body Mass Index (BMI) within the 18.5-30 kg/m2 range, to ensure a representative sample of the population
* Recent mammography and gynecological examination (within the last year) confirming the absence of breast or reproductive system diseases

Exclusion Criteria:

* Contraindications to hormone therapy, including a history of suspected or diagnosed malignancy
* Use of hormonal treatments or products derived from soybeans or cod liver oil within the last 12 months
* Allergies to soybeans or cod liver oil
* Engagement in professional athletic activities
* Current use of medications that may interact with study supplements, including but not limited to sulfonamides, methotrexate, triamterene, sulfasalazine, phenytoin, anxiolytics, antidepressants, as well as daily chemicals, multivitamins, aspirin, or painkillers
* Use of alternative herbal remedies for vasomotor symptoms within the past month
* Participation in another investigational program involving interventions outside of routine clinical practice within the last 6 months
* Presence of uncontrolled hypertension or diabetes, or a significant psychiatric condition that could interfere with study participation
* History of serious cardiovascular diseases, including myocardial infarction or stroke

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2023-07-18 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Change in the Menopause Rating Scale (MRS) score | 90 days
  Each symptom is rated on a scale from 0 (no complaints) to 4 (severe symptoms), leading to a total MRS score that ranges from 0 to 44

SECONDARY OUTCOMES:
Follicle-Stimulating Hormone (FSH) change | 90 days
Estradiol change | 90 days
Number of any adverse events | 90 days
  any reported adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Center of New Medical Technologies, Novosibirsk, Novosibisk Region, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pokushalov E, Ponomarenko A, Garcia C, Kasimova L, Pak I, Shrainer E, Romanova A, Kudlay D, Johnson M, Miller R. Assessing the combined effects of Black Cohosh, Soy Isoflavones, and SDG Lignans on menopausal symptoms: a randomized, double-blind, placebo-controlled clinical trial. Eur J Nutr. 2025 Mar 25;64(3):138. doi: 10.1007/s00394-025-03588-y. PMID 40131516